CLINICAL TRIAL: NCT00071227
Title: Pilot Study of Intravitreal Injection of Triamcinolone Acetonide Formulation for Retinal Vascular Disorders
Brief Title: Eye Injections of Triamcinolone Acetonide for Retinal Blood Vessel Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040013; 04-EI-0013
Record Dates: First submitted 2003-10-15; First posted 2003-10-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Macular Degeneration; Retinal Vein Occlusion
Keywords: Age Related Macular Degeneration; Macular Edema; Inflammation; Choroidal Neovascularization; CRVO; Diabetic Retinopathy; Age Related Macular Edema; AMD
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion; Macular Edema; Inflammation; Choroidal Neovascularization; Diabetic Retinopathy | interventions — Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide (TAC-PF)

SUMMARY:
This study will evaluate the safety and effectiveness of a new formulation of triamcinolone acetonide for the treatment of retinal blood vessel disorders. Triamcinolone is a steroid drug that decreases inflammation and scarring and is routinely used to treat eye inflammation or swelling. The commercially available form of this drug is associated with potentially harmful side effects thought to be due to preservatives in the preparation. This study will use a formulation that does not contain these potentially harmful preservatives. Preliminary findings from other studies suggest that injection of steroids in the eye can reduce retinal thickening and improve vision. However, they may also cause mild discomfort and lead to vision-threatening conditions. The effects of the drug on the conditions under study in this protocol are not known.

Patients with the following conditions involving disorders of retinal blood vessels may be eligible for this study:

* Choroidal neovascularization associated with age-related macular degeneration (50 years of age and older)
* Macular edema associated with retinal vein occlusion (18 years of age and older)
* Diabetic macular edema ((18 years of age and older)

Participants undergo the following tests and procedures:

* Medical history and physical examination
* Eye examination to assess visual acuity (eye chart test) and eye pressure, and to examine pupils, lens, retina and eye movements. The pupils will be dilated with drops for this examination.
* Fluorescein angiography to evaluate the eye's blood vessels. A yellow dye is injected into an arm vein and travels to the blood vessels in the eyes. Pictures of the retina are taken using a camera that flashes a blue light into the eye. The pictures show if any dye has leaked from the vessels into the retina, indicating possible blood vessel abnormality.
* Indocyanine green angiography to identify feeder vessels that may be supplying abnormal blood vessels. This procedure is similar to fluorescein angiography, but uses a green dye and flashes an invisible light.
* Optical coherence tomography to measure retinal thickness. This test shines a light into the eye and produces cross-sectional pictures of the retina. These measurements are repeated during the study to determine if retinal thickening is getting better or worse, or staying the same.
* Stereoscopic color fundus photography to examine the back of the eye. The pupils are dilated with eye drops to allow examination and photography of the back of the eye.
* Triamcinolone acetonide injection to treat the eye. A numbing eye drop, an antibiotic eye drop, and an injected antibiotic are put in the eye before triamcinolone acetonide is injected into the eye's vitreous (jelly-like substance inside the eye). After the injection, the patient lies on his or her back for 30 minutes. An antibiotic eye ointment is used for 2 days following treatment.
* Blood tests to measure liver and kidney function.

Patients return to the clinic for follow-up visits 1, 4, and 7 days, and 1 month after the first treatment. Patients whose condition does not improve after 3 months do not receive any more injections, but return for eye examinations at least once a year for 3 years. Patients whose condition improves with treatment return for follow-up visits 6 and 9 months after the first injection and then every 6 months for 2 more years. At each visit, a determination is made whether another injection is needed. After each repeat injection, patients return for follow-up visits at 1, 4, and 7 days after the injection.

DETAILED DESCRIPTION:
The use of intravitreal injections of corticosteroid (triamcinolone acetonide) appears to be a promising treatment for a variety of ocular diseases associated with inflammation. To date, the only drug available, 'Kenalog-40 Injection' produced by Bristol Myers Squibb, has not been formulated for intraocular use. This formulation when used intraocularly has been associated with cases of non-bacterial endophthalmitis, which is thought to be due to the presence of benzyl alcohol and/or polysorbate 80. Both are suspected irritants.

The purpose of this study is to evaluate the safety of a novel preservative-free formulation of triamcinolone acetonide (TAC-PF) at four dosage levels.

The study will be an open-label, single-masked, randomized Phase I study that will investigate the safety and potential efficacy of the new formulation of TAC-PF. Sixteen participants with retinal vascular disease will be randomly assigned to receive via intravitreal injection at one of 4 dose levels (1 mg, 4 mg, 8 mg, or 16 mg) of TAC-PF. Depending on a participant's response, injections may be repeated at up to 3 month intervals. Participants will be followed for 3 years.

The primary outcome will be an assessment of post-injection intraocular toxicity related events including increased inflammation, increased intraocular pressure, significant decreases in BCVA, cataract formation, retinal detachment, and intraocular hemorrhage. The secondary outcomes will be an improvement of 15 letters in best-corrected visual acuity (BCVA, ETDRS) from baseline to year 3, and decreases in retinal thickening and area of leakage.

ELIGIBILITY:
* INCLUSION CRITERIA - GENERAL:

All participants must:

1. Understand and sign the informed consent.
2. Must have visual acuity in the fellow eye the same or better than the study eye.
3. Have BCVA worse than 20/80 in the study eye.
4. Have sufficiently clear ocular media to permit good quality retinal photographs and angiography to allow assessment of the macular area according to standard clinical practice.
5. Be willing to use reliable forms of birth control during the study period.
6. Be able to comply with the study requirements.

INCLUSION CRITERIA - DISEASE-SPECIFIC:

Participants with neovascular AMD:

1. Have a diagnosis of AMD defined by the presence of drusen larger than 63 micrometers, in at least one eye.
2. Must be at least 50 years of age.
3. Have the presence of choroidal neovascularization under the fovea determined by the investigator and defined as any one of the following fluorescein angiographic (FA) features:

   1. Early stippled hyperfluorescence of flat retinal pigment epithelium with ill-defined boundary and little or mild leakage in the late frames of the fluorescein.
   2. Irregular elevation of the retinal pigment epithelium that does not exhibit discrete or bright hyperfluorescence in the early transit phase of the angiogram. Stippled hyperfluorescence may be present. Late frames may show persistent fluorescein staining or leakage within a sensory retinal detachment overlying this area.
   3. Late phase leakage of undetermined source with leakage at the level of the retinal pigment epithelium in the late frames of the angiogram in which the source of the late leakage cannot be determined from earlier-phase frames of the angiogram.
   4. A well-demarcated area of bright hyperfluorscence in the early phase of the angiogram with leakage through the mid- and late- phase frames which obscures the boundaries of the area.

Participants with central retinal vein occlusion:

1. Have macular edema in the study eye secondary to CRVO.
2. Must be at least 18 years of age.

Participants with diabetic macular edema:

1. Have clinically significant macular edema in the study eye secondary to diabetic retinpathy.
2. Must be at least 18 years of age.
3. Must have documented hemoglobin A1C of 12% or less within one month of baseline.

EXCLUSION CRITERIA - GENERAL:

All participants must not:

1. Have intraocular pressure greater than 25 or history suggesting glaucoma (e.g., history of the diagnosis of glaucoma, past or present use of medications to control intraocular pressure, or disc/nerve fiber layer defects suggestive of glaucoma) or glaucomatous visual field defects as documented by Goldmann or Humphrey perimetry taken within 6 months to qualification.
2. Be allergic to iodine or iodine-containing dyes.
3. Be allergic to fluorescein dyes.
4. Have medical conditions that make consistent follow-up over the treatment period unlikely (e.g., stroke, severe MI, or terminal carcinoma).
5. Be currently using or be likely to need systemic or ocular medications known to be toxic to the lens, retina, or optic nerve, such as:

   1. Deferoxamine
   2. Chloroquine/Hydroxychloroquine (Plaquenil)
   3. Tamoxifen
   4. Phenothiazines
   5. Ethambutol
6. Have a positive urine pregnancy test (for women of childbearing potential).
7. Have concurrent administration of other experimental therapies for the present disease.
8. Have any contraindication to performing the necessary diagnostic procedures.
9. Have a history of or current acute ocular or periocular infection (including any history of ocular herpes zoster or simplex).
10. Have had any major intraocular surgical procedure within one month of enrollment.
11. Have used ocular or systemic steroids or used steroid-containing inhalers or nasal sprays for more than 6 days a month, on average, or any regular use of pills containing steroids.
12. Have a known history of untoward complications from corticosteroid therapy, including elevated intraocular pressure in response to topical or periocular corticosteroids.
13. Have a history of other antiangiogenic treatment of concomitant administration of other therapies for the present disease.

EXCLUSION CRITERIA - DISEASE SPECIFIC:

Participants with Neovascular AMD must not:

1. Have any feeder vessels as seen on the high-speed ICG.
2. Have choroidal neovascularization (CNV) in the study eye, associated with other ocular diseases such as pathologic myopia, ocular histoplasmosis, or posterior uveitis.
3. Have geographic atrophy under the fovea in the study eye.
4. Have decreased vision, in the study eye, due to retinal disease not attributable to CNV, such as nonexudative forms of ARM, geographic atrophy, inherited retinal dystrophy, uveitis, or epiretinal membrane.
5. Have fibrosis, hemorrhage, pigment epithelial detachments, or other hypofluorescent lesions obscuring greater than 50% of the CNV lesion.

Participants with Central Retinal Vein Occlusion must not:

1. Have choroidal neovascularization.
2. Have had pan retinal laser photocoagulation within three months of randomization.

Participants with Diabetic Macular Edema must not:

1. Have had cataract surgery within six months of randomization.
2. Have had laser photocoagulation, either focal or scatter treatment, within three months of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2003-10-15; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Arvas S, Ocakoglu O, Ozkan S. The capillary blood flow in ischaemic type central retinal vein occlusion: the effect of laser photocoagulation. Acta Ophthalmol Scand. 2002 Oct;80(5):490-4. doi: 10.1034/j.1600-0420.2002.800506.x. PMID 12390159